CLINICAL TRIAL: NCT03130309
Title: Survival Rates of Atients Wearing a Mobile Unicompartimental Knee Prosthesis for the Past 10 Years
Brief Title: Results of a Mobile Unicompartimental Knee Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6756
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2017-04

CONDITIONS: Knee Replacement
Keywords: Knee; Replacement; Mobile-bearing; unicompartmental prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The unicompartmental knee prosthesis has become a routine procedure. Survival rate of over 90% after 10 years are generally reported. However, complications and reoperation may still occur for many reasons, and some of them may be related to component design: loosening (tibial above), polyethylene wear, knee stiffness, ligamentous instability, etc ... . Therefore, new designs can, at least in theory, improve the results of conventional models.

In this study, the investigators want to compare retrospectively data concerning survival rates of patients wearing unicompartmental knee prosthesis with mobile plate for over 10 years, with the ones published in the literature for conventional fixed-bearing prostheses and mobile-bearing prostheses

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients wearing unicompartmental knee prosthesis with mobile plate for over 10 years

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wearing unicompartmental knee prosthesis with mobile plate for over 10 years
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Compare retrospectively data concerning survival rates of patients wearingunicompartmental knee prosthesis with mobile plate for over 10 years, with the ones published in the literature for conventional fixed and mobile bearing prosthesis. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Centre de Chirurgie Orthopédique et de la Main (CCOM), Strasbourg, France

IPD SHARING:
Plan to Share IPD: No